CLINICAL TRIAL: NCT06821464
Title: Safety, Tolerability and Pharmacokinetics of HRS-9813 After Multiple Oral Administration in Healthy Subjects-A Phase I Clinical Study
Brief Title: A Trial of HRS-9813 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9813-102
Record Dates: First submitted 2025-02-05; First posted 2025-02-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis/Progressive Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): Low dose
  Interventions: Drug: HRS-9813
- Treatment group B (Experimental): High dose
  Interventions: Drug: HRS-9813

INTERVENTIONS:
Drug: HRS-9813 — Initial dose to planned dose（low dose）
  Arms: Treatment group A
Drug: HRS-9813 — Initial dose to planned dose（high dose）
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the safety and pharmacokinetics of HRS-9813 after multiple oral administration in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the start of activities related to this trial, and be able to fully understand the procedures, methods, contents and possible adverse reactions of this trial, and be willing to strictly abide by the clinical trial protocol to complete this trial.
2. Aged 18-45 years (inclusive), healthy male or female;
3. Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI): 19-26 kg/m2 (inclusive), body mass index (BMI) = weight (kg)/(height/100)2 (m2);
4. Physical examination, vital signs, 12-lead electrocardiogram, chest anteroposterior and lateral radiographs, abdominal ultrasound and laboratory tests during the screening and baseline periods were normal, or slightly abnormal but clinically insignificant as determined by the researchers;
5. Female subjects with fertility and male subjects whose partners are women of childbearing age have taken contraceptive measures within 2 weeks before signing the informed consent form, and are willing to abstain from sex or agree to contraception from the signing of the informed consent form until the end of the follow-up period (non-drug contraception is required during the trial, see Section 13.1.2 for details), and have no plans to have children or donate sperm/eggs.

Exclusion Criteria:

-

The following diseases or treatment history:

1. Any serious clinical diseases such as urinary system, circulatory system, endocrine system, nervous system, digestive system, respiratory system, blood system, immune system, mental and metabolic disorders in the past or currently, or any other diseases that the investigators judge may interfere with the results of the trial, such as intestinal diseases (including irritable bowel syndrome) and urinary tract infection/stones, etc.;
2. History of malignant tumors (cancers that have been confirmed to have been cured or relieved for ≥5 years, except for radically resected basal cell or squamous cell skin cancer, cervical cancer in situ and resected colon polyps);
3. Any conditions or diseases that affect the absorption, metabolism and/or excretion of the study drug;
4. Severe infection, severe trauma or major surgery within 3 months before the screening period or baseline period; or plan to undergo surgery during the trial;
5. Have used any drug in the 2 weeks before the screening or baseline period (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, dietary supplements, vitamin A and its derivatives, etc., excluding other conventional vitamins and occasional use of acetaminophen), or still within 5 half-lives of the drug during the screening or baseline period (whichever is longer); plan to use non-test drugs during the trial;
6. Participated in clinical trials of any other drugs or medical devices within 3 months before the screening or baseline period or planned to participate in the study period, or still within 5 half-lives of the drug during the screening or baseline period (whichever is longer);

   Any of the following examinations during screening meet the following criteria:
7. During the screening or baseline period, sitting systolic blood pressure <90 mmHg or sitting diastolic blood pressure <60 mmHg;
8. During the screening or baseline period, orthostatic hypotension occurs (retest within 15 minutes to confirm);
9. During the screening or baseline period, abnormal and clinically significant 12-lead electrocardiogram results, male QTcB>450ms, female QTcB>460ms;
10. During the screening or baseline period, serum creatinine exceeding the upper limit of normal (ULN);
11. During the screening or baseline period, eGFR < 70 mL/min/1.73m2 (calculated using the MDRD formula, eGFR (mL/min/1.73m2) = 175×(serum creatinine/88.4)-1.234×age-0.179×(0.79 female), where serum creatinine units are μmol/L);
12. During the screening or baseline period, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding 1.2 times ULN, or total bilirubin exceeding 1.5 times ULN;
13. During the screening period, any one of the following items is positive: hepatitis B virus surface antigen (HBsAg), human immunodeficiency virus antibody, syphilis spirochete antibody or hepatitis C virus antibody;

    General situation:
14. Pregnant or lactating women, or positive pregnancy test results during the screening period/baseline period;
15. History of blood donation or severe blood loss (blood loss ≥400 mL) within 8 weeks before the screening period or baseline period, or have received blood transfusion within 4 weeks before the screening period or baseline period; or intend to donate blood during the trial;
16. Have been vaccinated within 2 weeks before the screening period or baseline period or plan to be vaccinated during the trial;
17. History of smoking (average daily smoking >5 cigarettes) within 4 weeks before the screening period or baseline period, or cannot stop using any tobacco products during the trial;
18. Average daily alcohol intake exceeds 15 g (15 g alcohol is equivalent to 450 mL beer, 150 mL of wine or about 50mL of low-alcohol liquor), or cannot abstain from alcohol during the trial; or positive alcohol breath test at baseline;
19. History of drug abuse or drug dependence before the screening period or baseline period; or positive urine drug test at baseline;
20. Drink excessive amounts of tea, coffee or caffeinated beverages (more than 8 cups per day, 250 mL per cup) within 6 months before the screening period or baseline period;
21. Have consumed special foods (such as grapefruit, grapefruit juice or foods/beverages containing grapefruit juice, chocolate, tobacco, alcohol, caffeinated foods or beverages) within 48 hours before the baseline period;
22. Have special dietary requirements and cannot follow a unified diet;
23. Have difficulty swallowing, difficulty in venous blood collection, or physical conditions that cannot withstand intensive blood collection;
24. Other situations in which the researcher determines that the subject is not suitable for participating in this trial, including but not limited to the following: any physical or psychological disease or condition that may increase the risk of the trial, affect the subject's compliance with the protocol, or affect the subject's completion of the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Safety outcomes: Incidence and severity of AEs. | Day -14 to Day 22

SECONDARY OUTCOMES:
Area under the drug-time curve | Day 1 to Day 22
Area under the steady-state drug-time curve within the dosing interval | Day 1 to Day 22
Peak concentration | Day 1 to Day 22
Time to peak | Day 1 to Day 22
Half-life | Day 1 to Day 22
Apparent clearance | Day 1 to Day 22
Apparent volume of distribution | Day 1 to Day 22
Steady-state trough concentration | Day 1 to Day 22
Steady-state peak concentration[ | Day 1 to Day 22
Accumulation ratio (Racc) | Day 1 to Day 22
Proportion of subjects experiencing hypotension during the study | Day 1 to Day 22

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided